CLINICAL TRIAL: NCT02577614
Title: Factor VIII Inhibitor Bypass Activity (FEIBA) for the Reduction of Transfusion in Cardiac Surgery: A Randomized Double Blind Placebo Controlled Pilot Trial
Brief Title: FEIBA and Use of Blood Products in Cardiac Surgery
Acronym: FEIBA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Miriam Treggiari, Clinical Research Director, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11975
Record Dates: First submitted 2015-09-24; First posted 2015-10-16 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Cardiovascular Disease
Keywords: Cardiopulmonary Bypass; Aortic Valve Repair; Coronary Re-Implantation; Deep Hypothermic Circulatory Arrest; Factor VIII Inhibitor Bypass Activity; Transfusion
MeSH Terms: conditions — Cardiovascular Diseases | interventions — anti-inhibitor coagulant complex; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FEIBA (Experimental): Single dose of commercially available FEIBA
  Interventions: Drug: FEIBA
- Normal Saline (Placebo Comparator): Single dose of NaCl 0.9%
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: FEIBA — Administration of FEIBA after cardiopulmonary bypass
  Other Names: Anti-Inhibitor Coagulant Complex
  Arms: FEIBA
Drug: Normal Saline — Administration of placebo after cardiopulmonary bypass
  Other Names: NaCl 0.9%
  Arms: Normal Saline

SUMMARY:
The purpose of this pilot study is to evaluate the feasibility of the prophylactic administration of Factor VIII Inhibitor Bypass Activity (FEIBA) at termination of cardiopulmonary bypass (CPB) period. Specifically, the proposed study is designed to demonstrate the potential role of FEIBA administration in reducing the need for allogeneic transfusion to treat refractory coagulopathy in high risk patients.

DETAILED DESCRIPTION:
Factor eight inhibitor bypassing activity (FEIBA) is currently approved for use in this country for the treatment of patients with Hemophilia and inhibitors at a dose of 50-100 units/kg. There is a large body of evidence demonstrating the safety and efficacy of FEIBA for Hemophilia patients with inhibitor and has a theoretical advantage compared to current blood product transfusion methods, as it replenishes multiple depleted factors that are lost with prolonged exposure to CPB.

This pilot study is a single center, randomized, double-blinded, placebo controlled trial assessing the feasibility and safety of factor eight inhibitor bypass activity (FEIBA) in patients undergoing major cardiovascular surgery requiring prolonged CPB. The study population will consist of adult patients undergoing elective cardiac surgery at OHSU. Twelve participants will randomly assigned to receive FEIBA or placebo during their surgical procedure.

Patients will be followed to review for adverse events while in the ICU, and up to four weeks after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Elective aortic or aortic valve procedures, coronary re-implantation (Bentall) with cardiopulmonary bypass, and/or deep hypothermic circulatory arrest.
* Written informed consent

Exclusion Criteria:

* Contraindications to the administration of FIEBA or known anaphylactic or severe hypersensitivity reactions to FEIBA or any of its components
* Disseminated intravascular coagulation (DIC)
* Acute thrombosis or embolism, including myocardial infarction
* Pregnant women
* Decisionally impaired adults
* Prisoners
* Expressed unwillingness or are otherwise deemed unable to provide written informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Volume of blood products transfused (mL) | 30 days
  -Cumulative volume of blood products transfused, defined as the volume in mL of packed red blood cells, fresh frozen plasma, and platelets, after the administration of the study drug (mL)

SECONDARY OUTCOMES:
Number of thrombotic or thromboembolic events | 30 days
  - thrombotic or thromboembolic events are defined as any event of deep venous thrombosis, pulmonary embolism, stroke, or MI
Number of patients with post-operative bleeding requiring surgical hemostasis | 30 days
Duration of post-operative ventilation, ICU and hospital length of stay | 30 days
Number of deaths | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Sera VA, Stevens AE, Song HK, Rodriguez VM, Tibayan FA, Treggiari MM. Factor VIII inhibitor bypass activity (FEIBA) for the reduction of transfusion in cardiac surgery: a randomized, double-blind, placebo-controlled, pilot trial. Pilot Feasibility Stud. 2021 Jul 2;7(1):137. doi: 10.1186/s40814-021-00873-5. PMID 34215339